CLINICAL TRIAL: NCT00220272
Title: A Phase II, Randomized, Multicenter, Multinational, Double-Blind, Placebo-Controlled, Study of the Effect of SR57667B on Dopaminergic Nigro-Striatal Function Assessed by 18F-Dopa PET Imaging in Outpatients With Early Parkinson's Disease
Brief Title: Study of the Effect of SR57667B on 18F-Dopa PET Imaging in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT5288
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; 5-fluorodopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR57667B

SUMMARY:
* The primary objective is to study the effect of SR57667B at the dose of 4 mg/d on progression of dopaminergic nigro-striatal lesions assessed by 18F-Dopa PET imaging.
* Secondary objectives are to assess the effect of SR57667B on symptomatic decline in patients with early PD, to assess the safety/tolerability of SR57667B in patients with early PD and to document plasma concentrations of SR57667 in patients with early PD.

DETAILED DESCRIPTION:
Multinational, multicenter, randomized, parallel-group, double-blind, phase II study.Randomization stratified on the dopaminergic treatment, in two strata: treatment by levodopa or dopamine agonist.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients.
* Age >=35 years at screening.
* Diagnosis of Parkinson's syndrome, on at least two of the three key Parkinson's symptoms, i.e. resting tremor, bradykinesia and rigidity.
* Duration of the disease of less than 3 years since diagnosis.
* Modified Hoehn and Yahr stage <= 2.5.
* Patient optimized on monotherapy by levodopa or a dopamine agonist·
* Generally healthy and ambulatory.
* Patient has given his informed written consent and is capable of following study procedures.

Exclusion Criteria:

* Any indication of forms of parkinsonism other than PD.
* Severe resting tremor. Presence of either dyskinesia, fluctuations, or loss of postural reflexes·
* Treatment with amantadine, anticholinergics, catechol-o-methyltransferase (COMT ) inhibitors, selegiline, dopamine receptor antagonists, catecholamine depleters, indirect dopamine agonists or alphamethyldopa. Electroconvulsive therapy (ECT).Use of CYP3A4 strong, and moderate inducers or inhibitors. Participation in another clinical trial with an investigational drug within two months prior to randomization.
* Dementia, uncontrolled depression, psychotic disorder. History of substance-related disorders including alcohol or other substance use disorders.
* Females of child bearing potential.
* Evidence (detected by history, physical examination and/or laboratory/ECG tests) of any clinically significant or unstable medical disorder that could interfere with the patient's participation in the clinical trial; interfere with the absorption, metabolism or excretion of the study medication; or interfere with the evaluation of the study drug. Alterations of laboratory tests or ECG findings of potential clinical significance.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2004-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change in average (left and right) putamen 18F-Dopa influx constant (Ki) from baseline to two year 18F-Dopa PET

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Remy, MD, Study Chair — Service Hospitalier Frédéric Joliot, CEA, Orsay France
Locations (7):
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com